CLINICAL TRIAL: NCT02679950
Title: Understanding the Molecular and Genetic Differences Between GCT at the Time of the Initial Diagnosis and at Late Relapse
Brief Title: Understanding the Molecular and Genetic Differences Between Germ Cell Tumor at the Time of the Initial Diagnosis and at Late Relapse
Status: Completed | Type: Observational
Sponsor: Nasser Hanna (Other)
Responsible Party: Sponsor-Investigator, Nasser Hanna, Associate Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Other Study IDs: IUSCC-0540
Record Dates: First submitted 2015-11-09; First posted 2016-02-11 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Neoplasms, Germ Cell and Embryonal
Keywords: Next generation genome sequencing; Late relapse; Genetic profiles
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Initial diagnosis: The initial diagnosis only cohort will include 3 patients with germ cell tumor (GCT) who meet the inclusion criteria and have adequate tissue samples available in storage at the Pathology Department. One prospective blood and one tissue sample will be collected from each patient in this cohort. Tissue samples will come from the orchiectomy or virgin retro-peritoneal lymph node dissection (RPLND) that was done at initial diagnosis.
  Interventions: Genetic: Next generation genome sequencing
- Late relapse: The late relapse cohort will include 3 patients with late relapse germ cell tumor (GCT) who meet the inclusion criteria and have adequate tissue samples available in storage at the Pathology Department. One prospective blood and two tissue samples will be collected from each patient in this cohort. Tissue samples will come from the orchiectomy or virgin retro-peritoneal lymph node dissection (RPLND) that was done at initial diagnosis and the other will come from the site of late relapse.
  Patients in this cohort will have biopsies at the site of late relapse as part of their routine cancer treatment. No biopsies will be performed specifically for the purposes of this study. Tissue from the site of late relapse will also be requested from the Pathology Department.
  Interventions: Genetic: Next generation genome sequencing

INTERVENTIONS:
Genetic: Next generation genome sequencing — DNA will be extracted from each sample and assayed.

SUMMARY:
The current proposal is a pilot study. The Investigators plan to use next generation genome sequencing (NGGS) to define the molecular and genetic profiles of 3 cases of germ cell tumor (GCT) (with a component of yolk sac tumor) at the time of the initial diagnosis and 3 cases of late relapse GCT's, which are characterized by yolk sac tumor (and AFP secreting) predominant disease.

Investigators seek to demonstrate the feasibility of obtaining tissue biopsies (either archived or new biopsy) and utilization of NGGS in studying the molecular and genetic relationships between GCT's (with a component of yolk sac tumor) at the time of diagnosis and GCT's at the time of late relapse. This study will also provide preliminary information on genetic alterations, which may be a hypothesis for generating another study.

DETAILED DESCRIPTION:
This study will examine two cohorts:

1. The initial diagnosis only cohort will include 3 patients with GCT who meet the inclusion criteria and have adequate tissue samples available in storage at the Pathology Department. One prospective blood and one tissue sample will be collected from each patient in this cohort. Tissue samples will come from the orchiectomy or virgin retro-peritoneal lymph node dissection (RPLND) that was done at initial diagnosis.
2. The late relapse cohort will include 3 patients with late relapse GCT who meet the inclusion criteria and have adequate tissue samples available in storage at the Pathology Department. One prospective blood and two tissue samples will be collected from each patient in this cohort. Tissue samples will come from the orchiectomy or virgin RPLND that was done at initial diagnosis and the other will come from the site of late relapse.

Patients in this cohort will have biopsies at the site of late relapse as part of their routine cancer treatment. No biopsies will be performed specifically for the purposes of this study. Tissue from the site of late relapse will also be requested from the Pathology Department.

One tube of blood will be collected from each subject during a routine clinical visit at baseline when a blood draw is already being done.

In summary, a total of 15 samples will be evaluated on this study. Consent for the use of tissue and blood collected for the purposes of this study will be obtained prior to any study procedures. Subjects who do not have adequate tissue samples available will be replaced.

ELIGIBILITY:
Eligible patients will have:

1. Germ cell tumor (GCT) (with a component of yolk sac tumor) at the time of the initial diagnosis or a late relapsed GCT (for the purposes of this study, late relapse will be defined as relapse > 2 years from the initial treatment of GCT).
2. Adequate tumor specimens available from the initial orchiectomy specimen or virgin retro-peritoneal lymph node dissection (RPLND).
3. Adequate tumor specimens available from any site of recurrent disease for patients accrued in the "late relapse" cohort.
4. Tumor specimens collected prior to start of chemotherapy in the "late relapse" cohort.
5. Age > 18 years
6. Willing to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with germ cell tumor (GCT) (with a component of yolk sac tumor) at the time of the initial diagnosis or a late relapsed GCT.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
Compare genomic profiles of curable germ cell tumors with non curable germ cell tumors | 1 year
  Collection of tissue and blood samples from 6 patients for genomic testing

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, MD, Principal Investigator — Indiana University School of Medicine, Indiana University Simon Cancer Center
Locations (2):
- United States (2):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana